CLINICAL TRIAL: NCT00228891
Title: Effects of Pulsatile Insulin Delivery on Peripheral Diabetic Neuropathy
Brief Title: Effects of Pulsatile Insulin Delivery on Diabetic Neuropathy in Patients With Types 1 and 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other); Global Infusions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H09-66 NEU1; MH42900 and MH01386
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, With Complications
Keywords: Pulsatile intravenous insulin; Oral carbohydrate loading; Respiratory Quotients; Hypoglycemia; Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Complications; Hypoglycemia; Diabetic Neuropathies | interventions — Insulin, Regular, Human; Insulin Aspart

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Patients with diagnosed diabetic neuropathy will receive objective baseline testing and follow up testing every six months after the start of Pulsatile intravenous insulin therapy to monitor and assess diabetic neuropathy.
  Interventions: Procedure: Effect of Pulsatile IV Insulin on diabetic neuropathy
- 1 (Placebo Comparator): Control patients with diabetic neuropathy will receive objective testing at baseline and every six months to compare and measure results with patients who are receiving pulsatile intravenous insulin therapy.
  Interventions: Procedure: Effect of Pulsatile IV insulin on diabetic neuropathy

INTERVENTIONS:
Procedure: Effect of Pulsatile IV insulin on diabetic neuropathy — Control patients with diagnosed diabetic neuropathy will have objective testing at baseline and every six months to compare and measure results to patients receiving pulsatile intravenous insulin therapy.
  Arms: 1
Procedure: Effect of Pulsatile IV Insulin on diabetic neuropathy — Patients diagnosed with diabetic neuropathy will be treated with pulsatile intravenous insulin on a weekly basis. Patient's Endocrinologist will determine the dosage of intravenous insulin to be given each week based upon the patient's response and insulin resistance.
  Other Names: Humulog, Humulin, Novolog,
  Arms: 2

SUMMARY:
Diabetic neuropathy is a progressive complication causing serious problems in 25-40% of diabetic patients. Anecdotal reports have indicated improvement with pulsatile IV insulin in patients otherwise resistant to all conventional therapies. Significant complications produce painful peripheral dysesthesias, loss of sensation and gastroparesis. This study is designed to test the effectiveness of pulsatile insulin delivery on diabetic neuropathy.

DETAILED DESCRIPTION:
Diabetic neuropathy (DN) is a progressive complication causing serious problems in 25%-40% of diabetic patients. Significant complications produce painful peripheral dysesthesias, loss of sensation, and gastroparesis. DN may affect the peripheral motor and sensory nerves in addition to the autonomic nervous system (1-3). Treatment strategies for patients with DN have generally concentrated on pain relief, without addressing the underlying pathophysiology of the disease (4). Anecdotal reports from patients treated with pulsatile insulin for other complications suggest that this treatment may show efficacy in patients with DN. This study is designed to compare patients with DN who receive pulsatile insulin with a control group.

Pulses of IV insulin encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose insulin pulses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent measuring of glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions. The insulin pulses are delivered over 1-hour periods with a 1-hour rest period between each session. Three treatments are given during each treatment day.

The respiratory quotient (RQ) is a measurement of CO2 exhaled and O2 inhaled and is proportionate to the fuel sources being used by the body, primarily the liver over short periods of time. The higher the RQ, the more glucose and less alternative fuel sources are being utilized. Following the RQ change helps determine the effectiveness of physiological insulin administration in increasing anabolic functions in diabetic individuals. By improving the body's glucose metabolism and thereby causing beneficial effects of anabolic factors, the possibility of serious complications can be decreased. In addition the use of oral carbohydrate at the same time along with the physiologic insulin administration stimulates the appropriate gut hormones which augment this effect, a response which cannot be duplicated with intravenous glucose. The purpose of our studies is to determine whether the physiologic administration of insulin along with the augmenting effect of oral carbohydrates will normalize metabolism in diabetic patients and correlate with an improvement in their manifestations of diabetic neuropathy.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 30 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05.

1. Tesfaye S, Chaturvedi N, Eaton SEM, Ward JD, Manes C, Ionescu-Tirgoviste C, Witte DR, Fuller JH, Vascular Risk factors and Diabetic Neuropathy N Engl J Med 352:341-50, 2005.
2. Neuropathy Trust, Diabetic Neuropathy:Prevalence, www.neurocentre.com.
3. Potter PJ, Maryniak O, Yamorski R, Jones IC, Incidence of Peripheral Neuropathy in the Contralateral Limb of Persons with Unilateral Amputation due to Diabetes, Journal of Rehabilitation Research and Development 35:335-39, 1998.
4. Goldstein DJ, Lu Y, Detke MJ, Lee TC, Iyengan , Duloxetine versus Placebo in Patients with Painful Diabetic Neuropathy, Pain 116:109-18, 2005.

ELIGIBILITY:
Inclusion Criteria:

* The researchers will include up to 500 patients both male and female between the ages of 20 and 90 diagnosed with type 1 or type 2 diabetes mellitus.
* All patients were diagnosed by their endocrinologists as having diabetic neuropathy
* All patients had failed conventional treatment for diabetic neuropathy
* Taking oral agents and/or insulin for diabetic control
* Under an Endocrinologists supervision for their diabetes management. Endocrinologist must assess and approve patient for participation in this study
* Ability to swallow without difficulty
* Ability to commit to the weekly time requirements associated with the study

Exclusion Criteria:

* Other causes of complications not related to diabetes
* Lack of intravenous access
* Pregnancy
* Alcohol abuse, drug addiction or the use of illegal drugs
* Positive HIV
* Inability to breathe into machine for respiratory quotients

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Measure the stabilization or reduction of the decline of diabetic neuropathy by pt questionnaires and diagnostic tests | Measure the stabilization and reduction of complications associated with diabetic neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, PhD, Principal Investigator — Florida Atlantic University
Locations (1):
- Florida Atlantic University Center for Complex Systems and Brain Sciences, Boca Raton, Florida, United States

REFERENCES:
- [Background] Gill G, Moulik P. Mortality and diabetic neuropathy. Diabet Med. 2005 Sep;22(9):1289. doi: 10.1111/j.1464-5491.2005.01729.x. No abstract available. PMID 16108870
- [Background] Moghtaderi A, Bakhshipour A, Rashidi H. Validation of Michigan neuropathy screening instrument for diabetic peripheral neuropathy. Clin Neurol Neurosurg. 2006 Jul;108(5):477-81. doi: 10.1016/j.clineuro.2005.08.003. Epub 2005 Sep 16. PMID 16150538
- [Background] Tesfaye S, Chaturvedi N, Eaton SE, Ward JD, Manes C, Ionescu-Tirgoviste C, Witte DR, Fuller JH; EURODIAB Prospective Complications Study Group. Vascular risk factors and diabetic neuropathy. N Engl J Med. 2005 Jan 27;352(4):341-50. doi: 10.1056/NEJMoa032782. PMID 15673800
- [Background] Potter PJ, Maryniak O, Yaworski R, Jones IC. Incidence of peripheral neuropathy in the contralateral limb of persons with unilateral amputation due to diabetes. J Rehabil Res Dev. 1998 Jul;35(3):335-9. PMID 9704317
- [Background] Goldstein DJ, Lu Y, Detke MJ, Lee TC, Iyengar S. Duloxetine vs. placebo in patients with painful diabetic neuropathy. Pain. 2005 Jul;116(1-2):109-18. doi: 10.1016/j.pain.2005.03.029. PMID 15927394